CLINICAL TRIAL: NCT01623050
Title: SinuSys Patency of Maxillary Sinus Ostia Study
Brief Title: Safety and Performance of the SinuSys Dilation System for Dilation of the Maxillary Sinus Ostium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SinuSys Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS-005
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SinuSys Dilation System (Experimental): Maxillary Sinus Dilation
  Interventions: Device: SinuSys Dilation System

INTERVENTIONS:
Device: SinuSys Dilation System — Sinuplasty

SUMMARY:
The purpose of this study is to assess safety and performance of the SinuSys Dilation System for dilation of the maxillary sinus ostium.

DETAILED DESCRIPTION:
A multicenter, single-arm, prospective study conducted to assess the safety and effectiveness of a new osmotically-driven, low-pressure expansion device for dilation of maxillary sinus ostia in patients with (CRS) Chronic Rhinosinusitis

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of chronic maxillary sinusitis

Exclusion Criteria:

* Previous antrostomy
* Sinonasal tumours
* Cystic fibrosis
* History of facial trauma that distorts sinus anatomy and precludes access to the maxillary sinus
* Pregnant or breastfeeding females
* Currently participating in another drug or device study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Catalano, MD, Principal Investigator — St Elizabeth Medical Center; Amin Javer, MD, Principal Investigator — St. Paul's Hospital
Locations (5):
- United States (3):
  - Valley ENT, Tucson, Arizona
  - Palo Alto Medical Foundation, Palo Alto, California
  - St. Elizabeth Medical Center, Boston, Massachusetts
- St. Paul's Hospital, ENT Department, Vancouver, British Columbia, Canada
- Charing Cross Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SinuSys Dilation System
Started | 36
Treated | 34
Completed | 27
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Population: 36 patients were enrolled; 2 patients withdrew consent prior to treatment.
Arm/Group | SinuSys Dilation System
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (16.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21
  Canada | 12
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Patency of Treated Area
Time Frame: Immediately post procedure
Population: Number of osita treated
Measure: Number; unit: percentage of ostia treated
Units Other Than Participants: Ostia
Arm/Group | SinuSys Dilation System
Number analyzed (Participants) | 34
Number analyzed (Ostia) | 59
percentage of ostia treated | 95

2. Secondary Outcome: Patency of Treated Area
Description: Maxillary Sinus Ostia Patency of 33 patients analyzed.
Time Frame: 3 months
Population: One patient was lost to follow up
Measure: Number; unit: percentage of ostia patent
Units Other Than Participants: Ostia
Arm/Group | SinuSys Dilation System
Number analyzed (Participants) | 33
Number analyzed (Ostia) | 55
percentage of ostia patent | 93

3. Secondary Outcome: Number of Participants With Device-related Adverse Events as a Measure of Safety
Time Frame: 3 months
Measure: Number; unit: number of participants
Arm/Group | SinuSys Dilation System
Number analyzed (Participants) | 34
number of participants | 0

4. Secondary Outcome: Patency of Treated Area
Description: Maxillary Sinus Ostia Patency of 29 patients analyzed.
Time Frame: 6 months
Population: 5 patients were lost to follow up
Measure: Number; unit: percentage of ostia patent
Units Other Than Participants: Ostia
Arm/Group | SinuSys Dilation System
Number analyzed (Participants) | 29
Number analyzed (Ostia) | 47
percentage of ostia patent | 91

5. Secondary Outcome: Patency of Treated Area
Description: Maxillary Sinus Ostia of 27 patients analyzed.
Time Frame: 12 months
Population: 7 patients were lost to follow up
Measure: Number; unit: percentage of ostia patent
Units Other Than Participants: Ostia
Arm/Group | SinuSys Dilation System
Number analyzed (Participants) | 27
Number analyzed (Ostia) | 45
percentage of ostia patent | 93

ADVERSE EVENTS:
Description: Only device related adverse events collected
Arm/Group | SinuSys Dilation System
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less